CLINICAL TRIAL: NCT04471779
Title: The IDEAL Study: Information About Alzheimer's Disease for Latinos in New York City
Brief Title: Information About Alzheimer's Disease for Latinos in New York City
Acronym: IDEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Ruth Ottman, Professor of Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AAAR8269; R01AG062528 (NIH)
Record Dates: First submitted 2020-07-09; First posted 2020-07-15 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-07

CONDITIONS: Alzheimer Disease
Keywords: Latinos; New York (NY); Genetics
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: The investigators estimate that 2171 people will participate in the Baseline Survey, of whom 400 will be randomized and included in the follow-up study. Half of those in the follow-up study will be randomized to receive information about their risk of Alzheimer's disease based on Latino ethnicity, family history, and APOE genotype, and half will be randomized to receive information about their risk based on ethnicity and family history alone.
Who Masked: Outcomes Assessor
Masking Description: Persons conducting follow-up surveys via computer-assisted telephone interviews will be masked with respect to participant randomization group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Disclosure (Experimental): Participants will be given information about their risk of Alzheimer's disease based on Latino ethnicity, family history of Alzheimer's disease, and their APOE genotype.
  Interventions: Other: Disclosure of APOE genotype
- Non-disclosure (No Intervention): Participants will be given information about their risk of Alzheimer's disease based on Latino ethnicity and family history of Alzheimer's disease alone.

INTERVENTIONS:
Other: Disclosure of APOE genotype — Information about risk of Alzheimer's disease will be given to participants based on their APOE genotypes, in addition to Latino ethnicity and family history.
  Arms: Disclosure

SUMMARY:
This study will assess the psychosocial and behavioral impacts of receiving Alzheimer's disease genetic risk assessment incorporating APOE genotypes among Latinos in northern Manhattan. The investigators will conduct a longitudinal, community-based study with a mixed methods design. Participants will be randomized to learn about their lifetime risk of late-onset Alzheimer's disease (AD) based either on (a) Latino ethnicity and family history alone (genotype nondisclosure group), or (b) the same factors plus APOE genotype (genotype disclosure group). Responses will be evaluated at 6 weeks, 9 months, and 15 months after risk assessment. In the quantitative component of the study, the investigators will assess psychosocial outcomes, memory test performance, and health-related behaviors. In the qualitative component of the study, the investigators will investigate the lived experience of receiving personal AD risk information, using a stress and coping theoretical framework.

DETAILED DESCRIPTION:
Apolipoprotein E (APOE) is the strongest genetic predictor of risk for late-onset Alzheimer's disease (AD). Given the high level of interest in genetic testing, the demand for predictive testing for APOE will surely increase. Improved understanding of the impacts of testing, sources of variability in response, and inclusion of diverse samples are critical for informing methods to promote safe and effective disclosure of AD genetic risk information.

As with other diseases, previous research on AD, a devastating and incurable illness, has found little significant or sustained distress in response to genetic susceptibility testing for APOE, even among persons who learn they are at elevated risk. These surprising findings, which run counter to the experience of many clinicians, may be related to limitations in the methods of previous studies. Most previous studies primarily enrolled well-educated Caucasians with a family history, who were strongly motivated to pursue genetic risk information. Further, most studies assessed impacts primarily through standardized measures of depression and anxiety, which may not capture the kinds of distress experienced or coping strategies that might blunt or mask distress. Qualitative research shows that receipt of genetic information can have important psychosocial effects not well captured through standardized measures. Also, in one study, people with a high-risk gene test for APOE performed worse on memory tests if they were informed about the results than if they were not informed, suggesting that other impact measures are needed.

Another important limitation of prior work is that it has lacked representation of ethnic minority groups. Latinos are the second largest U.S. ethnic group, comprising about 18% of the population, yet no previous study has investigated the impacts of receiving AD genetic risk information among Latinos. While AD incidence rates may vary among Latino subgroups, data from the Washington Heights-Inwood Columbia Aging Project (WHICAP), a study in northern Manhattan, indicate that they are about twice as high among Caribbean Hispanics (primarily Dominicans) as among persons of European ancestry.

In this study, the investigators will improve understanding of the impacts of receiving personal AD genetic risk information and the factors that influence adjustment to such information among Latinos who live in the same communities studied in WHICAP.

ELIGIBILITY:
Inclusion Criteria:

* self-identified as Latino or Hispanic
* age 40-64 years
* current residence in target neighborhoods: Washington Heights, Inwood, Hamilton Heights, Central Harlem, East Harlem, Morningside Heights, Manhattanville, or Striver's Row, New York

Exclusion Criteria:

* does not self-identify as Latino
* does not reside in target neighborhoods
* not in applicable age range
* has Alzheimer's disease
* previously tested for APOE
* has a family history consistent with autosomal dominant, early onset Alzheimer's disease
* has a positive screen for suicidality in Baseline Survey (any response other than "not at all" to PHQ-9 item, "thoughts that you would be better off dead or of hurting yourself in some way")

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 374 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2025-10-03 (Actual); Study Completion 2025-10-03 (Actual)

PRIMARY OUTCOMES:
Impact of Genetic Testing in AD (IGT-AD) | 6 weeks after risk evaluation
  16-item scale that assesses the impact of test result disclosure across both distress and positive domains. The scale will be modified to anchor it to "risk assessment" rather than genetic test results to enable it to be used in both disclosure groups. Each item scored 0 (never), 1 (rarely) 3 (sometimes) 5 (often). Values are summed; higher total indicates worse outcome (greater adverse impact). Scale range: 0-80.
Impact of Genetic Testing in AD (IGT-AD) | 9 months after risk evaluation
  16-item scale that assesses the impact of test result disclosure across both distress and positive domains. The scale will be modified to anchor it to "risk assessment" rather than genetic test results to enable it to be used in both disclosure groups. Each item scored 0 (never), 1 (rarely) 3 (sometimes) 5 (often). Values are summed; higher total indicates worse outcome (greater adverse impact). Scale range: 0-80.
Impact of Genetic Testing in AD (IGT-AD) | 15 months after risk evaluation
  16-item scale that assesses the impact of test result disclosure across both distress and positive domains. The scale will be modified to anchor it to "risk assessment" rather than genetic test results to enable it to be used in both disclosure groups. Each item scored 0 (never), 1 (rarely) 3 (sometimes) 5 (often). Values are summed; higher total indicates worse outcome (greater adverse impact). Scale range: 0-80.
Impact of Event Scale-Revised | 6 weeks after risk evaluation
  22-item scale to assess subjective distress caused by traumatic events. Each item scored on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Subscales can be calculated for Intrusion, Avoidance, and Hyperarousal. The authors recommend using means instead of summed scores; higher mean score indicates worse outcome (greater impact). Scale range: 0-4.
Impact of Event Scale-Revised | 9 months after risk evaluation
  22-item scale to assess subjective distress caused by traumatic events. Each item scored on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Subscales can be calculated for Intrusion, Avoidance, and Hyperarousal. The authors recommend using means instead of summed scores; higher mean score indicates worse outcome (greater impact). Scale range: 0-4.
Impact of Event Scale-Revised | 15 months after risk evaluation
  22-item scale to assess subjective distress caused by traumatic events. Each item scored on a 5-point scale ranging from 0 ("not at all") to 4 ("extremely"). Subscales can be calculated for Intrusion, Avoidance, and Hyperarousal. The authors recommend using means instead of summed scores; higher mean score indicates worse outcome (greater impact). Scale range: 0-4.
Change in Score on the Brief Test of Adult Cognition by Telephone (BTACT) | Baseline and 6 weeks after risk evaluation
  15-20 minute test of cognitive differences in normal aging. Composite score (the average of standardized z-scores for six measures: immediate memory, delayed memory, working memory, verbal fluency, speed, and reasoning. Lower scores indicate worse outcome (worse memory performance). Range of scale values: -1 to +1.
Change in Score on the Brief Test of Adult Cognition by Telephone (BTACT) | Baseline and 9 months after risk evaluation
  15-20 minute test of cognitive differences in normal aging. Composite score (the average of standardized z-scores for six measures: immediate memory, delayed memory, working memory, verbal fluency, speed, and reasoning. Lower scores indicate worse outcome (worse memory performance). Range of scale values: -1 to +1.
Change in Score on the Brief Test of Adult Cognition by Telephone (BTACT) | Baseline and 15 months after risk evaluation
  15-20 minute test of cognitive differences in normal aging. Composite score (the average of standardized z-scores for six measures: immediate memory, delayed memory, working memory, verbal fluency, speed, and reasoning. Lower scores indicate worse outcome (worse memory performance). Range of scale values: -1 to +1.
Change in Score on the Metamemory in Adulthood Questionnaire-Revised | Baseline and 6 weeks after risk evaluation
  20-item test of subjective memory. Each item measured on a 5-point Likert scale from 1 (agree strongly) to 5 (disagree strongly). Lower scores indicate worse outcome (worse subjective memory functioning and more decline in memory across time). Scale range: 20-100.
Change in Score on the Metamemory in Adulthood Questionnaire-Revised | Baseline and 9 months after risk evaluation
  20-item test of subjective memory. Each item measured on a 5-point Likert scale from 1 (agree strongly) to 5 (disagree strongly). Lower scores indicate worse outcome (worse subjective memory functioning and more decline in memory across time). Scale range: 20-100.
Change in Score on the Metamemory in Adulthood Questionnaire-Revised | Baseline and 15 months after risk evaluation
  20-item test of subjective memory. Each item measured on a 5-point Likert scale from 1 (agree strongly) to 5 (disagree strongly). Lower scores indicate worse outcome (worse subjective memory functioning and more decline in memory across time). Scale range: 20-100.

SECONDARY OUTCOMES:
Change in Score on Patient Health Questionnaire-9 (PHQ-9) | Baseline and 6 weeks after risk evaluation
  9-item screen for depressive symptoms. Each item rated by the frequency with which symptoms were experienced during the preceding 2 weeks (0-3, with 3 most frequent). Scores are summed; higher total indicates worse outcome (more depressive symptoms). Scale range: 0-27.
Change in Score on Patient Health Questionnaire-9 (PHQ-9) | Baseline and 9 months after risk evaluation
  9-item screen for depressive symptoms. Each item rated by the frequency with which symptoms were experienced during the preceding 2 weeks (0-3, with 3 most frequent). Scores are summed; higher total indicates worse outcome (more depressive symptoms). Scale range: 0-27.
Change in Score on Patient Health Questionnaire-9 (PHQ-9) | Baseline and 15 months after risk evaluation
  9-item screen for depressive symptoms. Each item rated by the frequency with which symptoms were experienced during the preceding 2 weeks (0-3, with 3 most frequent). Scores are summed; higher total indicates worse outcome (more depressive symptoms). Scale range: 0-27.
Change in Score on the General Anxiety Disorder-7 (GAD-7) | Baseline and 6 weeks after risk evaluation
  7-item screen for anxiety symptoms. Each item rated by self-reported severity of a given symptom over the past 2 weeks from 0 (not at all) to 3 (nearly every day). Higher total score indicates worse outcome (more anxiety symptoms). Scale range: 0-21.
Change in Score on the General Anxiety Disorder-7 (GAD-7) | Baseline and 9 months after risk evaluation
  7-item screen for anxiety symptoms. Each item rated by self-reported severity of a given symptom over the past 2 weeks from 0 (not at all) to 3 (nearly every day). Higher total score indicates worse outcome (more anxiety symptoms). Scale range: 0-21.
Change in Score on the General Anxiety Disorder-7 (GAD-7) | Baseline and 15 months after risk evaluation
  7-item screen for anxiety symptoms. Each item rated by self-reported severity of a given symptom over the past 2 weeks from 0 (not at all) to 3 (nearly every day). Higher total score indicates worse outcome (more anxiety symptoms). Scale range: 0-21.
Change in Perceived Threat of AD | Baseline and 6 weeks after risk evaluation
  7-item scale to assess perceived threat of developing Alzheimer's disease. Each item rated on 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Scores are summed; higher scores indicate worse outcome (more threat). Scale range: 7-35.
Change in Perceived Threat of AD | Baseline and 9 months after risk evaluation
  7-item scale to assess perceived threat of developing Alzheimer's disease. Each item rated on 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Scores are summed; higher scores indicate worse outcome (more threat). Scale range: 7-35.
Change in Perceived Threat of AD | Baseline and 15 months after risk evaluation
  7-item scale to assess perceived threat of developing Alzheimer's disease. Each item rated on 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Scores are summed; higher scores indicate worse outcome (more threat). Scale range: 7-35.
Health-related behavior changes | 6 weeks after risk evaluation
  22 items, with each item answered yes (1) or no (0). Total value greater than 0 indicates better outcome (the participant made a change in diet, exercise, or medications/vitamins in response to receiving genetic information).
Health-related behavior changes | 9 months after risk evaluation
  22 items, with each item answered yes (1) or no (0). Total value greater than 0 indicates better outcome (the participant made a change in diet, exercise, or medications/vitamins in response to receiving genetic information).
Health-related behavior changes | 15 months after risk evaluation
  22 items, with each item answered yes (1) or no (0). Total value greater than 0 indicates better outcome (the participant made a change in diet, exercise, or medications/vitamins in response to receiving genetic information).
Recall/understanding of results | 6 weeks after risk evaluation
  5 questions will be asked to assess recall of results, each of which is answered correctly or incorrectly. Outcome is the total number of correct answers (0 thru 5). Higher score indicates better outcome.
Recall/understanding of results | 9 months after risk evaluation
  5 questions will be asked to assess recall of results, each of which is answered correctly or incorrectly. Outcome is the total number of correct answers (0 thru 5). Higher score indicates better outcome.
Recall/understanding of results | 15 months after risk evaluation
  5 questions will be asked to assess recall of results, each of which is answered correctly or incorrectly. Outcome is the total number of correct answers (0 thru 5). Higher score indicates better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Ottman, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from surveys collected in the study will be made available from the PIs, after acceptance for publication of the primary analyses of the survey data, to qualified researchers who sign a data user agreement as described below. The investigators will provide documentation of all survey data (variable names, variable formats, variable and value labels) to accompany the data, and will share the actual survey instruments upon request. Because interview transcripts can be highly identifying, they will not be shared. However, the codebooks and interview guides will be available from the PIs, after acceptance for publication of the primary analyses of the interviews, to qualified users as described below.
Supporting Information: Study Protocol, Analytic Code
Time Frame: After acceptance for publication of the primary analyses of the study.
Access Criteria: Data will be available to users only under a data user agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.
  Requests for data must be in writing and addressed to the co-PIs. We will create a data request form that will include investigator affiliation, contact information and a brief description of the project, including specific aims, study design, characteristics of the data requested, and analysis plans. Applications for data use will be reviewed by the co-PIs and a data use committee composed of the other co-investigators. Approval will be contingent upon institutional review board (IRB) approval for the proposed data analysis from the institution of the investigator requesting the data.

REFERENCES:
- [Background] Molinuevo JL, Pintor L, Peri JM, Lleo A, Oliva R, Marcos T, Blesa R. Emotional reactions to predictive testing in Alzheimer's disease and other inherited dementias. Am J Alzheimers Dis Other Demen. 2005 Jul-Aug;20(4):233-8. doi: 10.1177/153331750502000408. PMID 16136847
- [Background] Heshka JT, Palleschi C, Howley H, Wilson B, Wells PS. A systematic review of perceived risks, psychological and behavioral impacts of genetic testing. Genet Med. 2008 Jan;10(1):19-32. doi: 10.1097/GIM.0b013e31815f524f. PMID 18197053
- [Background] Green RC, Roberts JS, Cupples LA, Relkin NR, Whitehouse PJ, Brown T, Eckert SL, Butson M, Sadovnick AD, Quaid KA, Chen C, Cook-Deegan R, Farrer LA; REVEAL Study Group. Disclosure of APOE genotype for risk of Alzheimer's disease. N Engl J Med. 2009 Jul 16;361(3):245-54. doi: 10.1056/NEJMoa0809578. PMID 19605829
- [Background] Bemelmans SA, Tromp K, Bunnik EM, Milne RJ, Badger S, Brayne C, Schermer MH, Richard E. Psychological, behavioral and social effects of disclosing Alzheimer's disease biomarkers to research participants: a systematic review. Alzheimers Res Ther. 2016 Nov 10;8(1):46. doi: 10.1186/s13195-016-0212-z. PMID 27832826
- [Background] Vos J, van Asperen CJ, Oosterwijk JC, Menko FH, Collee MJ, Gomez Garcia E, Tibben A. The counselees' self-reported request for psychological help in genetic counseling for hereditary breast/ovarian cancer: not only psychopathology matters. Psychooncology. 2013 Apr;22(4):902-10. doi: 10.1002/pon.3081. Epub 2012 Jun 27. PMID 22740372
- [Background] Gooding HC, Linnenbringer EL, Burack J, Roberts JS, Green RC, Biesecker BB. Genetic susceptibility testing for Alzheimer disease: motivation to obtain information and control as precursors to coping with increased risk. Patient Educ Couns. 2006 Dec;64(1-3):259-67. doi: 10.1016/j.pec.2006.03.002. Epub 2006 Jul 21. PMID 16860524
- [Background] Zallen DT. "Well, good luck with that": reactions to learning of increased genetic risk for Alzheimer disease. Genet Med. 2018 Nov;20(11):1462-1467. doi: 10.1038/gim.2018.13. Epub 2018 Mar 8. PMID 29517767
- [Background] Lineweaver TT, Bondi MW, Galasko D, Salmon DP. Effect of knowledge of APOE genotype on subjective and objective memory performance in healthy older adults. Am J Psychiatry. 2014 Feb;171(2):201-8. doi: 10.1176/appi.ajp.2013.12121590. PMID 24170170
- [Background] Aviles-Santa ML, Heintzman J, Lindberg NM, Guerrero-Preston R, Ramos K, Abraido-Lanza AL, Bull J, Falcon A, McBurnie MA, Moy E, Papanicolaou G, Pina IL, Popovic J, Suglia SF, Vazquez MA. Personalized medicine and Hispanic health: improving health outcomes and reducing health disparities - a National Heart, Lung, and Blood Institute workshop report. BMC Proc. 2017 Oct 3;11(Suppl 11):11. doi: 10.1186/s12919-017-0079-4. eCollection 2017. PMID 29149222
- [Background] Mehta KM, Yeo GW. Systematic review of dementia prevalence and incidence in United States race/ethnic populations. Alzheimers Dement. 2017 Jan;13(1):72-83. doi: 10.1016/j.jalz.2016.06.2360. Epub 2016 Sep 4. PMID 27599209
- [Background] Tang MX, Maestre G, Tsai WY, Liu XH, Feng L, Chung WY, Chun M, Schofield P, Stern Y, Tycko B, Mayeux R. Relative risk of Alzheimer disease and age-at-onset distributions, based on APOE genotypes among elderly African Americans, Caucasians, and Hispanics in New York City. Am J Hum Genet. 1996 Mar;58(3):574-84. PMID 8644717
- [Background] Tang MX, Stern Y, Marder K, Bell K, Gurland B, Lantigua R, Andrews H, Feng L, Tycko B, Mayeux R. The APOE-epsilon4 allele and the risk of Alzheimer disease among African Americans, whites, and Hispanics. JAMA. 1998 Mar 11;279(10):751-5. doi: 10.1001/jama.279.10.751. PMID 9508150
- [Background] Gurland BJ, Wilder DE, Lantigua R, Stern Y, Chen J, Killeffer EH, Mayeux R. Rates of dementia in three ethnoracial groups. Int J Geriatr Psychiatry. 1999 Jun;14(6):481-93. PMID 10398359
- [Background] Tang MX, Cross P, Andrews H, Jacobs DM, Small S, Bell K, Merchant C, Lantigua R, Costa R, Stern Y, Mayeux R. Incidence of AD in African-Americans, Caribbean Hispanics, and Caucasians in northern Manhattan. Neurology. 2001 Jan 9;56(1):49-56. doi: 10.1212/wnl.56.1.49. PMID 11148235
- [Background] Grubs RE, Parker LS, Hamilton R. Subtle psychosocial sequelae of genetic test results. Current Genetic Medicine Reports 2014;2:242-249.
- [Derived] Caban M, Tran E, Meng A, Wetmore JB, Ottman R, Siegel K. Planning for the future following receipt of Alzheimer's disease risk estimate among Latinos in New York City. J Alzheimers Dis. 2025 Oct;107(3):1226-1239. doi: 10.1177/13872877251365571. Epub 2025 Aug 8. PMID 40776633
- [Derived] Tran E, Caban M, Meng A, Wetmore JB, Ottman R, Siegel K. Knowledge and Beliefs About Medical and Non-Medical Interventions to Control Alzheimer's Disease Among Latinos in New York City. Int J Geriatr Psychiatry. 2025 Jul;40(7):e70128. doi: 10.1002/gps.70128. PMID 40627435
- [Derived] Meng A, Caban M, Tran E, Wetmore JB, Ottman R, Siegel K. Addressing Disparities in Alzheimer's Disease-Related Healthcare Through Understanding Factors Contributing to Perceived Vulnerability Among Latinos in Northern Manhattan: A Qualitative Report. J Racial Ethn Health Disparities. 2025 Apr 7:10.1007/s40615-025-02409-6. doi: 10.1007/s40615-025-02409-6. Online ahead of print. PMID 40195275